CLINICAL TRIAL: NCT03205787
Title: Red Clover Botanical Dietary Supplements - Metabolism and Safety in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Elena Barengolts, Principle Investigator, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2017-0436
Record Dates: First submitted 2017-06-29; First posted 2017-07-02 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Food-drug Interaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trifolium pratense (Experimental): Red clover extract; 2 gelatin capsules (398 mg extract) per day for 14 days
  Interventions: Dietary Supplement: Trifolium pratense

INTERVENTIONS:
Dietary Supplement: Trifolium pratense — Red Clover extract standardized to isoflavone content.
  Other Names: Red Clover

SUMMARY:
Human safety studies were carried out to test whether red clover botanical dietary supplements used by peri- and post-menopausal women are safe to use with Food and Drug Administration (FDA)-approved drugs. To test this, a red clover dietary supplement (previously tested in women at the University of Illinois at Chicago without any harmful effects) was given with four selected FDA-approved drugs to determine if the red clover supplement can increase or decrease how these medications are absorbed, metabolized and excreted by the human body. Preclinical studies predicted that the red clover supplement might affect the metabolism or break down of these probe drugs.

DETAILED DESCRIPTION:
At the start of a study, subjects were administered low doses of a mixture of four FDA-approved drugs (caffeine, tolbutamide, dextromethorphan, and alprazolam), and serial blood samples were drawn and analyzed for the concentration of each drug over time. Afterwards, participants took the red clover dietary supplement twice orally daily for 14 days to allow for potential inhibition or induction of drug metabolizing enzymes and transporters. Thereafter, the same drugs were taken again to obtain a second measure of drug concentrations in blood over time. Changes in the concentration-time curve values for each probe drug obtained before and after ingestion of the supplement were evaluated to determine if metabolism of the probe drugs was impacted by the red clover dietary supplement.

ELIGIBILITY:
Inclusion Criteria:

* healthy peri- and post-menopausal women ages 40 - 79
* non-smokers
* no-significant medical conditions as assessed by subject-reported medical history, physical examination and blood and urine chemistry screens
* no medical condition that requires chronic use of medication

Exclusion Criteria:

* known allergies or hypersensitivity to caffeine, dextromethorphan, sulfonylureas (tolbutamide), benzodiazepines, or red clover
* positive pregnancy test
* use of hormone therapy within 8 weeks of study initiation for oral agents, 4 weeks for transdermal or other topical agents
* use of caffeine products 7 days before study participation or during the study
* use of citrus products 7 days before study participation or during the study
* other prescription (with the exception of the Mirena® IUD) or non-prescription medicines within the 2 weeks prior to study initiation or during the study
* chronic diseases, such as inflammatory bowel disease, that could alter the absorption or metabolism of the probe substrates
* unwillingness to comply with study requirements
* current participation in another clinical trial
* CYP2D6 deficiency based on phenotyping at screening
* smoker
* red clover or soy intake (whether as a botanical dietary supplement, food, drink or otherwise) within the previous two weeks and during the study
* use of any dietary supplements within the last 2 weeks prior to study initiation and during the study
* extreme obesity (defined as >40 BMI)
* alcohol or drug abuse
* chronic diseases such as diabetes.

Ages: 40 Years to 79 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2020-04-29 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve (AUC) | baseline and 14 days
  Concentrations of probe drugs from blood draws at the conclusion of the 14-day intervention were used to calculate areas under the (extrapolated) concentration-time curve to determine any changes compared to pre-intervention.

SECONDARY OUTCOMES:
Apparent Clearance | baseline and 14 days
  Concentrations of probe drugs from blood draws at the conclusion of the 14-day intervention were used to calculate changes in apparent clearance of each probe drug compared to pre-intervention.
Peak Concentration | baseline and 14 days
  Concentrations of probe drugs from blood draws at the conclusion of the 14-day intervention were used to calculate changes in peak concentrations of probe drugs to compared to pre-intervention concentrations.
Time for Peak Concentration | baseline and 14 days
  Concentrations of probe drugs from blood draws at the conclusion of the 14-day intervention were used to calculate changes in time for peak concentration of probe drugs compared to pre-intervention concentrations.
Drug Half-life | baseline and 14 days
  Concentrations of probe drugs from blood draws at the end of the 14-day intervention were used to calculate half-lives of probe drugs to determine any changes compared to pre-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Richard vanBreemen, PhD, Study Director — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Muchiri RN, van Breemen RB. Single-Laboratory Validation of UHPLC-MS/MS Assays for Red Clover Isoflavones in Human Serum and Dietary Supplements. J AOAC Int. 2020 Jul 1;103(4):1160-1166. doi: 10.1093/jaoacint/qsaa033. PMID 33241325